CLINICAL TRIAL: NCT03028506
Title: Meal Composition and Frequency in Type 1 Diabetic Women and the Influence on Pre-prandial Blood Glucose Values and Fetal Weight.
Brief Title: Meal Composition and the Influence on Pre-prandial Blood Glucose Values
Status: Completed | Type: Observational
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Rosemary Catanzaro, RD, Principal Investigator, St. Louis University
Other Study IDs: 25217
Record Dates: First submitted 2017-01-19; First posted 2017-01-23 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Diabetes in Pregnancy
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Carbohydrate intake — By calculating carbohydrate amounts at meals and snacks, as well as classifying meals and snacks as high fat, the investigators will examine the correlation to higher preprandial blood glucose values and large for gestational age infants.

SUMMARY:
The purpose of the proposed study is to assess the distribution of carbohydrates and fat in the diet of women with type 1 diabetes during pregnancy. More specifically, it will look at the distribution of carbohydrate in the diet during weeks 29-32 of pregnancy. The carbohydrate distribution and fat content of the meal will be compared to maternal glucose control, preprandial glucose levels, and the percentile for weight of the infant at birth. In addition, each meal and snack will be classified as low-moderate fat or high fat.

DETAILED DESCRIPTION:
This is a retrospective chart review. Data will be collected on all patients seen whose blood sugar and food logs were at least 75% complete. By calculating carbohydrate amounts at meals and snacks, as well as classifying meals and snacks as high fat, we will examine the correlation to higher preprandial blood glucose values and large for gestational age infants. Preprandial glucose levels will be reviewed, questioning whether the biggest contributor is the composition of the previous meal or additional snacks between meals.

ELIGIBILITY:
Inclusion Criteria:

* Female, age 16-45, all ethnic groups,
* Type 1 diabetes
* Blood glucose logs at least 75% complete
* Food intake records during weeks 29-32 that are at least 75% complete

Exclusion Criteria:

* Maternal medical conditions:

  * Renal disease
  * Restrictive lung disease
  * Cyanotic heart disease (severe heart disease where mother is blue)
  * Antiphospholipid antibody syndrome
  * Collagen-vascular disease (lupus)
  * Substance use and abuse (drugs)
  * Multiple gestation
  * Genetic disorders
  * Severe malnutrition

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pregnant, all ethnic groups
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
large for gestational age infants | 1 year
  weight at birth

CONTACTS AND LOCATIONS:
Overall Officials: Rosemary Catanzaro, RD, Principal Investigator — St. Louis University

IPD SHARING:
Plan to Share IPD: No